CLINICAL TRIAL: NCT05421806
Title: A Cohort Study of Use of Doravirine (DOR) Based Regimens in Clinical Practice in Europe
Brief Title: A Cohort Study of Use of Doravirine (DOR) Based Regimens in Clinical Practice in Europe DoRavirine Europe Real World/
Acronym: DrEW
Status: Active, not recruiting | Type: Observational
Sponsor: NEAT ID Foundation (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: NEAT1010; NEAT 1010 (Other: NEAT ID)
Record Dates: First submitted 2022-06-10; First posted 2022-06-16 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: HIV I Infection
Keywords: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Cohort 1: 400 patients with no resistance mutations to DOR or NNRTIs.
- Cohort 2: Approximately 50 patients with resistance mutations to NNRTIs (other than DOR)
- Cohort 3: Approximately 50 patients with or without NNRTI mutations (including DOR)

SUMMARY:
Following the initiation of Doravirine (DOR) regimen among people living with HIV (PLWH), the study will aim to assess effectiveness, discontinuation, and resistance over the 12-month period.

Retrospective data from 500 patients is planned to be collected from 6 - 10 European sites. Cohort 1 : 400 patients, 100 treatment naïve and 300 virally suppressed patients switching from a 1st or second line treatment, Cohort 2: 50 patients with NNRTI mutations (other than DOR), Cohort 3: 50 patients with NNRTI mutations (including DOR).

The study will be conducted through collaboration with the NEAT ID Network, a well-established network of clinical sites across Europe.

ELIGIBILITY:
Inclusion Criteria:

* are HIV positive male or female
* are aged ≥18 years
* were prescribed and received at least one dose of DOR (without initial dose adjustment).
* have started/been switched to DOR for at least 12 months at time of data collection
* had a resistance genotype available before starting DOR

Cohort 1 Specific Inclusion Criteria

* had no evidence of DOR-associated resistance mutation
* were on DOR containing ART regimen that also contained 2 fully active nucleos(t)ides and patient had no documented NRTI resistance mutations to the two NRTIs in the combination.
* Patients who, at the time of initiation, were:

  1. Category 1: HIV treatment naïve OR
  2. Category 2: Virologically suppressed (HIV-1 RNA <50 copies/mL) for at least 6 months with no evidence of prior virological failure with agents of the NNRTI class

Patients in category 1 and 2 above who have NNRTI mutations that do not impact on DOR (K103N, Y181C, and G190A) using the Stanford algorithm (https://hivdb.stanford.edu/hivdb/by-mutations) can be included in this study.

Cohort 2 Specific Inclusion Criteria

* must have evidence of NNRTI associated resistance mutations (other than DOR) according to Stanford algorithm
* their DOR-containing ART will contain 2 NRTIs but will not include an INSTI and/or a bPI.
* had no documented resistance to the other drugs in the combination.
* Patients who, at the time of initiation, were:

  1. Category 1: HIV treatment naïve OR
  2. Category 2: Virologically suppressed (HIV-1 RNA <50 copies/mL) for at least 6 months

     Cohort 3 Specific Inclusion Criteria
* ART naïve or virologically suppressed (HIV-1 RNA <50 copies/mL) for at least 6 months at the time of DOR initiation

Exclusion Criteria:

* Patients with no documented resistance testing.
* Patients with no genotype available at DOR initiation
* Patients enrolled in DOR trials

Cohort 1 specific exclusion criteria

* Patients who have DOR as part of their fourth line or higher therapy
* Patients with prior virological failure with agents of the NNRTI class

Cohort 2 specific exclusion criteria

* Patients who have an INSTI and/or bPI in their DOR-containing therapy
* Patients who have NNRTI mutations that impact on DOR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-1 infected patients ≥ 18 years who were ART-naïve or virologically suppressed (VL < 50 copies for more than 6 months) and have been started/switched to DOR for at least 12 months at time of data collection.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-10-10 (Actual); Primary Completion 2026-03-06 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Proportion virologically suppressed patients at week 48 who have remained on DOR. | Week 48 after DOR initiation
  Proportion of patients, virologically suppressed/undetectable (<50 copies/mL) at week 48 who have remained on DOR.
Proportion of patients with virologic failure (Cohort 1 - treatment naive) | on or after week 48 after DOR initiation
  i. Two consecutive HIV RNA VL levels ≥50 copies/mL after reaching at HIV RNA < 50 copies/mL or ii. One HIV RNA VL level ≥50 copies/mL and DOR regimen is discontinued immediately or at next hospital visit, after reaching HIV RNA < 50 copies/mL
Proportion of patients with virologic failure (Cohort 2 - treatment suppressed) | up to 12 months after initiation of DOR
  i. Two consecutive HIV RNA VL levels ≥50 copies/mL after reaching at HIV RNA < 50 copies/mL or ii. One HIV RNA VL level ≥50 copies/mL and DOR regimen is discontinued immediately or at next hospital visit, after reaching HIV RNA < 50 copies/mL
Proportion of patients switched for reasons other than virological failure. | up to 12 months after initiation of DOR
  Proportion of patients switched at any time point for reasons other than virological failure.

SECONDARY OUTCOMES:
Proportion of patients with confirmed virologic failure, commonly used to make treatment related clinical decisions (Cohort 1 - treatment naive) | on or after week 48 after DOR initiation
  i. Two consecutive HIV RNA VL levels ≥200 copies/mL after reaching HIV RNA < 200 copies/mL or ii. One HIV RNA VL level ≥200 copies/mL and DOR regimen is discontinued immediately or at next hospital visit, after reaching HIV RNA < 200 copies/mL.
Proportion of patients with confirmed virologic failure, commonly used to make treatment related clinical decisions (Cohort 1 - treatment naive) | up to 12 months after initiation of DOR
  i. Two consecutive HIV RNA VL levels ≥200 copies/mL after reaching HIV RNA < 200 copies/mL or ii. One HIV RNA VL level ≥200 copies/mL and DOR regimen is discontinued immediately or at next hospital visit, after reaching HIV RNA < 200 copies/mL.
Estimated proportion of patients with low level viremia | up to 12 months after initiation of DOR
  Estimated proportion of patients with low level viremia (≥50-<200 copies/mL)
HIV resistance subtypes for patients with virologic failure | during the 12-month data collection period.
  HIV resistance mutations subtypes for all DOR treated patients with virologic failure

CONTACTS AND LOCATIONS:
Overall Officials: Anton Pozniak, Study Director — Chelsea and Westminster NHS Trust
Locations (19):
- Belgium (2):
  - Institute Of Tropical Medicine Antwerp, Antwerp
  - Saint-Pierre University Hospital, Brussels
- France (11):
  - Hospital Center University De Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - CHU Nantes University Hospital, Nantes
  - Hospital Center University De Nice, Nice
  - Bichat-Claude Bernard Hospital, Paris
  - Hopital Universitaire Pitie-Salpetriere, Paris
  - Hospital Saint Antoine, Paris
  - Lariboisière Hospital, Paris
  - Saint-Louis Hospital, Paris
  - St Louis Hospital, Paris
  - University Hospitals Pitié Salpêtrière, Paris
- Erasmus University Medical Center, Rotterdam, Netherlands
- Hospital Clínic de Barcelona, Barcelona, Spain
- United Kingdom (4):
  - Southmead Hospital, Bristol
  - Chelsea and Westminster Hospital, London
  - Guy's Hospital, London
  - Mortimer Market Center, Central and North West London NHS Trust, London

IPD SHARING:
Plan to Share IPD: No